CLINICAL TRIAL: NCT05510531
Title: A Study to Evaluate the Feasibility and Acceptability of a Diabetes Survival Skills + (DSS+) Training Intervention for Incarcerated Persons Transitioning to the Community (TTC)
Brief Title: Diabetes Survival Skills + (DSS+) Training Intervention for Incarcerated Persons Transitioning to the Community (TTC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: American Nurses Foundation (Other)
Responsible Party: Principal Investigator, Louise Reagan, Assistant Professor, University of Connecticut
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-066
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The proposed study will examine the feasibility, acceptability and preliminary efficacy measures of a quasi-experimental non-equivalent control group 6-week intervention study with repeated measures at baseline, 6 weeks, and 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Diabetes Survival Skills (DSS)Training (Experimental): Participants in the treatment group received a 6-session 1-hour weekly literacy tailored DSS education intervention.
  Interventions: Behavioral: Diabetes Survival Skills Training
- Control No intervention (No Intervention): Participants in the Control facility received the intervention upon completion of week twelve measurements.

INTERVENTIONS:
Behavioral: Diabetes Survival Skills Training — During the course of the DSS sessions, participants receive blood glucose logs, glucose meters; lancets, testing strips and demonstration insulin pens with injecting pillow will only be used in class. In summary, the DSS is focused on increasing knowledge, motivation, and self-efficacy and decreasing diabetes related distress, IMB components relevant to incarcerated persons and proximal to behavior change, through engagement, return demonstrations, skill practice, and positive reinforcement.
  Arms: Treatment Diabetes Survival Skills (DSS)Training

SUMMARY:
The purpose was to examine the feasibility and acceptability of a Diabetes Survival Skills intervention training with and without a support group for incarcerated persons transitioning to the community. Feasibility will include limited efficacy testing to examine the effect of the DSS+ intervention on diabetes knowledge, self-efficacy, outcome expectancies, and diabetes-related distress.

DETAILED DESCRIPTION:
Prison programs often lack efficacious diabetes self-management education (DSME)or skill-based programs to prepare citizens with diabetes when transitioning from a highly dependent secure environment to independent community living. There have been efforts to examine the effect of engaging incarcerated persons in blood glucose monitoring on glycemic control,11 but for the most part incarcerated persons or those recently released have not been included in decades of research involving community dwelling and ethnically diverse persons in numerous effective tailored and culturally relevant group/individual models of DSME for improving diabetes knowledge,12-14 self-care behavior (SCB),11,12,14 and stimulating participation in proactive risk reduction;16,17because incarcerated adults are considered a vulnerable population. These adults often have some cognitive dysfunction18 with lower than average prose, as well as decreased literacy across age, sex, and educational attainment, than those living in community households.19 With release into the community, these individuals undergo significant stress due to competing demands such as finding housing, and employment that can adversely affect DSM. It is unknown whether the evidence based DSME strategies used in the general community such as with discharge from the hospital to home are feasible, acceptable and effective for best supporting the transition of incarcerated persons in their continued DSM into the community. For example, one study reported prisoners, at seven days' post prison release, had higher rates of hospitalization for short-term diabetes complications and lower extremity amputations compared to matched controls.3 Interviews with recently released prisoners revealed significant stress post-release related to not knowing how and when to take insulin.20 In another study, respondents reported lack of knowledge regarding what foods to eat, how to control their blood sugar, take medications, or access health care. 21 At a minimum, incarcerated persons transitioning to the community have a critical need for DSS. Therefore, the purpose of this study is to evaluate the feasibility, acceptability and preliminary efficacy of implementing a 6 week DSS Training Intervention in the correctional setting 6-9months before incarcerated persons transition to the community.

Specific aims:

1. The primary aim is to evaluate feasibility of the experimental protocol: H1) Recruitment: 48 eligible persons will consent to participate in the study within 2 months. H2) Attendance/Attrition: 90% of enrolled participants will attend and complete the 6-session DSS Training. H3) Engagement: 75% of enrolled participants' will document responses to work-book questions, record blood glucose and if applicable associated diet or activity information. H4) Intervention implementation: The intervention will be delivered according to the DSS timeline (Figure1) and session outline. H5) Skill proficiency: Participants will return demonstrate how to use the blood glucose meter, insulin pen (as indicated), and blood glucose log, and other skills specific to DSS session 1-6.

The secondary aim is to elicit information about the participant's acceptability of the DSS intervention including perspective in participating in the intervention using focus groups.

3. The tertiary aim is to explore the preliminary efficacy and short term impact of the DSS Intervention on diabetes knowledge, outcome expectancies, emotional distress, and self-efficacy (Information-Motivation-Behavior Model [IMB]22,23 outcomes) at baseline, 6 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Eligible individuals:

* have Type 1 or 2 diabetes
* be male gender
* age 18 and older
* any race, or ethnicity
* be able to speak, and understand Englis
* within 6-9 months of being released from prison
* have a Connecticut Department of Corrections (CDOC) security and medical classification allowing participation in group sessions

Exclusion:

• none. See inclusion

Exclusion Criteria: none. See inclusion

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change in diabetes knowledge | Measured at Baseline and 6 and 12 weeks from baseline
  measured by Spoken knowledge for Low Literacy in Diabetes (SKILLD) , a 10-item scale that measures diabetes knowledge e.g. medication taking, blood glucose monitoring
Change in diabetes-related distress | Measured at Baseline and 6 and 12 weeks from baseline.
  Problem Areas in Diabetes Scale (PAID) measures diabetes-related distress.
Change in self-confidence for managing diabetes | Measured at Baseline and 6 and 12 weeks from baseline
  Self confidence in Diabetes Index(SCODI) Confidence Subscale 38 measures the degree of confidence the person has about his or her ability to perform specific self-care task and to persist in forming an action despite barriers
Change in outcome expectancy | Measured at Baseline and 6 and 12 weeks from baseline.
  Outcome Expectancy Questionaire(OEQ) measures a "person's perceptions of the consequences of performing diabetes self-care behavior

SECONDARY OUTCOMES:
Participants perspective of the intervention | Focus group interview performed between 8-12 weeks after the session/intervention is delivered.
  Focus groups to perspective about the overall quality of the program? Or how well did the program prepare you for transitioning to the community?

CONTACTS AND LOCATIONS:
Overall Officials: Louise Reagan, PhD, Principal Investigator — UCONN School of Nursing
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Todd S, Reagan L, Laguerre R. Health Literacy, Cognitive Impairment, and Diabetes Knowledge Among Incarcerated Persons Transitioning to the Community: Considerations for Intervention Development. J Forensic Nurs. 2023 Oct-Dec 01;19(4):262-270. doi: 10.1097/JFN.0000000000000396. Epub 2022 Apr 28. PMID 35482339
- [Result] Reagan L, Laguerre R, Todd S, Gallagher C. The Feasibility and Acceptability of a Diabetes Survival Skills Intervention for Persons Transitioning from Prison to the Community. J Racial Ethn Health Disparities. 2024 Apr;11(2):1014-1023. doi: 10.1007/s40615-023-01581-x. Epub 2023 May 8. PMID 37154888

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT05510531/Prot_SAP_ICF_000.pdf